CLINICAL TRIAL: NCT02082639
Title: Immunogenicity and Safety Study of GSK Biologicals' Human Papillomavirus (HPV) Vaccine (Cervarix™) (GSK-580299) When Co-administered With GSK Biologicals' Hepatitis A Vaccine (Havrix®) (GSK-208109) in Healthy Female Adolescents Aged 9-14 Years
Brief Title: Immunogenicity and Safety Study of GlaxoSmithKline (GSK) Biologicals' Human Papillomavirus Vaccine (Cervarix™) When Co-administered With GSK Biologicals' Hepatitis A Vaccine (Havrix®) in Healthy Female Adolescents Aged 9-14 Years
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Because the Russian Authorities already approved the 2-dose Cervarix™ schedule, the study was no longer needed for registration and hence it was cancelled.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 117099; 2012-004378-24 (EudraCT Number)
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-07

CONDITIONS: Infections, Papillomavirus
Keywords: Adolescents; Havrix; Immunogenicity; Cervarix; Safety
MeSH Terms: conditions — Papillomavirus Infections | interventions — human papillomavirus vaccine, L1 type 16, 18; Hepatitis A Vaccines

ARMS (3):
- HPV Group (Experimental): Subjects will receive two doses of HPV vaccine intramuscularly
  Interventions: Biological: Cervarix™
- HAV Group (Experimental): Subjects will receive two doses of HAV vaccine intramuscularly
  Interventions: Biological: Havrix
- HPV+HAV Group (Experimental): Subjects will receive two doses of both HPV and HAV vaccines intramuscularly
  Interventions: Biological: Cervarix™; Biological: Havrix

INTERVENTIONS:
Biological: Cervarix™ — 2 doses intramuscularly in the deltoid muscle of the non-dominant arm
  Arms: HPV Group; HPV+HAV Group
Biological: Havrix — 2 doses intramuscularly in the deltoid muscle of the dominant arm
  Arms: HAV Group; HPV+HAV Group

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of two doses of GSK Biologicals' HPV-16/18 L1 VLP AS04 vaccine when co-administered with GSK Biologicals' HAV vaccine according to 0, 6 month schedule, compared to the administration of either of these vaccines alone. The study will ascertain that the immune responses elicited to the two vaccines are not adversely impacted compared to when HPV-16/18 L1 VLP AS04 vaccine and HAV vaccine are administered alone.

ELIGIBILITY:
Inclusion Criteria:

* A female between, and including, 9 and 14 years of age at the time of the first vaccination.
* Subjects' parent(s)/Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject and informed assent obtained from the subject, if appropriate, prior to enrollment.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for two months after completion of the vaccination series.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period (up to Month 12).
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. Inhaled and topical steroids are allowed.
* Planned administration/administration of a vaccine not foreseen by the study protocol within the period starting 30 days before and 30 days after the first dose of vaccine with the exception of routine vaccines such as meningococcal, pertussis, inactivated influenza, diphtheria/tetanus and/or diphtheria/tetanus-containing vaccines up to 8 days before the first dose of study vaccine.
* Concurrently participating in another clinical study, at any time during the study period (up to Month 12), in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Previous vaccination against HPV or planned administration of any HPV vaccine other than that foreseen by the study protocol during the study period (up to Month 12).
* Previous administration of MPL or AS04 adjuvant.
* Previous vaccination against hepatitis A or planned administration of any hepatitis A vaccine other than that foreseen by the study protocol during the study period (up to Month 12).
* Cancer or autoimmune disease under treatment.
* History of hepatitis A infection.
* Known exposure to hepatitis A within the previous 6 weeks.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* Hypersensitivity to latex.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests, which in the opinion of the investigator preclude administration of the study vaccine.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period (up to Month 12).
* Acute disease and/or fever at the time of enrollment.

  * Fever is defined as temperature ≥ 37.0°C for oral, axillary or tympanic route. The preferred route for recording temperature in this study will be oral or axillary.

Ages: 9 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Anti-HPV-16/18 seroconversion status in the HPV group and the HPV+HAV group | One month after the second dose (Month 7)
Anti-HPV-16/18 antibody titres in the HPV group and the HPV+HAV group | One month after the second dose (Month 7)
Anti-HAV seroconversion status in the HPV+HAV group and the HAV group | One month after the second dose (Month 7)
Anti-HAV antibody titres in the HPV+HAV group and the HAV group | One month after the second dose (Month 7)

SECONDARY OUTCOMES:
Anti-HPV-16/18 seroconversion status in the HPV group and the HPV+HAV group | One month after the second dose (Month 7)
Anti-HPV-16/18 antibody titres in the HPV group and the HPV+HAV group | One month after the second dose (Month 7)
Anti-HAV seroconversion status in the HPV+HAV group and the HAV group | One month after the second dose (Month 7)
Anti-HAV antibody titres in the HPV+HAV group and the HAV group | One month after the second dose (Month 7)
Occurrence of any and Grade 3 solicited local symptoms (injection site pain, redness and swelling) in all study groups | During the 7-day period (Day 0-6) following each vaccination
Occurrence of any, Grade 3 and causally related to vaccination solicited general symptoms in all study groups | During the 7-day period (Day 0-6) following each vaccination
Occurrence of any, Grade 3 and causally related to vaccination unsolicited AEs in all study groups | During the 30-day period (Day 0-29) following any vaccination
Occurrence of any and causally related to vaccination serious adverse events (SAEs) in all groups | Throughout the active phase of the study (up to Month 7) and during the extended safety follow-up period (up to Month 12)
Occurrence of medically significant conditions (MSCs) in all groups | Throughout the active phase (up to Month 7) and during the extended safety follow-up period (up to Month 12)
Occurrence of potential immune-mediated diseases (pIMDs) in all groups | Throughout the active phase (up to Month 7) and during the extended safety follow-up period (up to Month 12)
Occurrence of pregnancies and pregnancy outcomes | During the entire study period (Month 0 - Month 12)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline